CLINICAL TRIAL: NCT02700815
Title: A Randomized, Controlled Multi-centre Parallel Group Study to Assess the Efficacy and Safety of Multiple Doses of a Topically Applied Combination Containing Diclofenac 2% + Capsaicin 0.075% (2 g Formulation Per Application; 2-times Daily for 5 Days) Compared to Placebo, as Well as to Diclofenac 2% and Capsaicin 0.075% in Patients With Acute Back or Neck Pain
Brief Title: Capsaicin + Diclofenac Gel in Acute Back Pain or Neck Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1358.1; 2015-000404-25 (EudraCT Number)
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Diclofenac; Capsaicin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Diclofenac and capsaicin (Experimental): Fixed dose combination
  Interventions: Drug: Diclofenac; Drug: Capsaicin
- Diclofenac (Active Comparator)
  Interventions: Drug: Diclofenac
- Capsaicin (Active Comparator)
  Interventions: Drug: Capsaicin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac
  Arms: Diclofenac; Diclofenac and capsaicin
Drug: Capsaicin
  Arms: Capsaicin; Diclofenac and capsaicin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This randomised, controlled multi-centre parallel group trial will assess the efficacy and tolerability of a topical formulation gel of the combination of diclofenac and capsaicin in comparison to gels with diclofenac alone, capsaicin alone, and placebo for the treatment of acute back pain or neck pain

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent at Visit 1 in accordance with Good Clinical Practice and local legislation
* Male or female patients >=18 years with current diagnosis of acute back pain or of neck pain for at least 24 hours, but less than 21 days
* Acute back pain or acute neck pain resulting in pain on movement (POM) >= 50 mm (Visual Analogue Scale 0-100) for at least one POM procedure out of 5 standardized procedures.
* Sensitivity to algometric pressure on the painful trigger point <= 25 N/cm2
* Women of childbearing potential must be ready and able to use highly effective methods of birth control

Exclusion criteria:

* History of 3 or more episodes of back or neck pain in the last 6 months excluding the current episode
* Surgery due to back or neck pain or rehabilitation due to back or neck pain in the last 12 months
* Back or neck pain that is attributable to any specific identifiable cause (e.g. disc prolapse, spondylolisthesis, osteomalacia, inflammatory arthritis, metabolic, neurological diseases or tumour)
* Trauma or strains of the back or neck muscles within the last 3 months
* Prior use within the last 3 days before Visit 1 or concomitant use of any anti-inflammatory drugs, heparinoids, muscle relaxants or analgesics. Long-acting glucocorticoids must have been discontinued 10 days before study entry. Spinal injections should have been discontinued in due time (investigator's judgement) before patient enrolment to allow complete wash-out of the active ingredient based on investigator's judgment
* Non-pharmacological treatment (physiotherapy, heat treatment (e.g. heat patch, hot water bottle), or massage, acupuncture, transcutaneous electrical nerve stimulation) or locally applied pharmacological product to the back or neck area 24 hours prior study entry and during the study period
* Known severe hepatocellular insufficiency, severe renal insufficiency or Gilbert's syndrome (Morbus Meulengracht)
* Any other medical condition that would interfere with efficacy and safety assessments based on investigator's judgement or any on-going clinical condition that would jeopardize patient's or site personnel's safety or study compliance based on investigator judgement.
* Known intolerance or hypersensitivity to the active ingredients or any excipient(s).
* Patients in whom attacks of asthma, bronchospasm, rhinitis or urticaria were precipitated by the intake of Acetyl salicylic acid (ASS) or other NSAIDs
* Irritated skin (based on investigator's judgement), skin wounds, eczema or open injuries at application site
* Negative experience in the past with heat treatments for muscle complaints
* Patient not able to understand and comply with trial requirements based on investigators judgement
* Alcohol or drug abuse
* Participation in a clinical trial within the previous 30 days or simultaneous participation in another clinical trial
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (18):
- Germany (14):
  - emovis GMBH, Berlin, Berlin
  - Synexus Clinical Research GmbH, Berlin
  - Synexus Clinical Research GmbH, Bochum
  - Sport- und Präventionsmedizinische Praxis, 50933 Köln, Cologne
  - Dünnwaldpraxis, Köln, Cologne
  - Praxis Dr. Steinebach, Essen, Essen
  - Praxis Dr. Schaefer, 45355 Essen, Essen
  - Unterfrintroper Hausarztzentrum, Essen
  - Synexus Clinical Research GmbH, Frankfurt
  - Praxis Dr. Pabst, Gilching, Gilching
  - Praxis Dr. Dahmen, 22415 Hamburg, Hamburg
  - Praxis Dr. Klein, Künzing, Künzing
  - Synexus Clinical Research GmbH, Leipzig
  - Anästhesiologie Rheinbach, Rheinbach
- Russia (4):
  - University Clinic of Headache, Private Practice, Moscow, Moscow
  - State Budget.Hlthcare Inst.City Outpatient dept #123,Therapy, Saint Petersburg
  - Medical Centre "Reavita", Therapy Dept., St. Petersburg, Saint Petersburg
  - St.Petersburg State Budget.Hlthcare Inst.City Outpat.dep#107, Saint Petersburg

REFERENCES:
- [Derived] Predel HG, Ebel-Bitoun C, Peil B, Weiser TW, Lange R. Efficacy and Safety of Diclofenac + Capsaicin Gel in Patients with Acute Back/Neck Pain: A Multicenter Randomized Controlled Study. Pain Ther. 2020 Jun;9(1):279-296. doi: 10.1007/s40122-020-00161-9. Epub 2020 Mar 27. PMID 32221866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, placebo and active treatment-controlled, double-blind, parallel group study. Out of 757 enrolled patients with acute back or neck pain, 746 were randomised and treated with 4 topical treatments administered twice daily for 4 to 7 days.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be entered to trial if any of the specific entry criteria were not met.
Groups:
- Placebo Gel: Patients were topically applied matching Placebo 2 gram (g) gel, twice daily with 12 ± 4 hours (h) between applications.
- Capsaicin (0.075%) Gel: Patients were topically applied Capsaicin 2 g gel (1.5 milligram (mg) Capsaicin), twice daily with 12 ± 4 hours (h) between applications.
- Diclofenac (2%) Gel: Patients were topically applied Diclofenac 2 g gel (40 milligram (mg) Diclofenac), twice daily with 12 ± 4 hours (h) between applications.
- Diclofenac (2%) +Capsaicin (0.075%) Gel: Patients were topically applied Diclofenac + Capsaicin 2 g gel (40 mg diclofenac, 1.5 mg capsaicin), twice daily with 12 ± 4 hours (h) between applications.
Period: Overall Study
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Started | 75 | 223 | 223 | 225
Completed | 74 | 216 | 219 | 218
Not Completed | 1 | 7 | 4 | 7
Not completed — Adverse Event | 0 | 6 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Refusal to continue medication | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All randomised patients who used at least 1 dose of study medication were included in the TS. Patients who received the wrong treatment were analysed within the planned (randomised) treatment group in the efficacy analysis and within the actual treatment group in the safety analysis (TS, as treated).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel | Total
Number analyzed (Participants) | 75 | 223 | 223 | 225 | 746
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of all patients included in the trial. Population: TS
  Years | 45.3 (14.78) | 43.2 (15.42) | 44.0 (15.96) | 44.2 (15.49) | 43.9 (15.52)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution of all patients included in the trial. Population: TS
  Participants
    Female | 44 | 128 | 136 | 136 | 444
    Male | 31 | 95 | 87 | 89 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of all patients included in the trial. Population: TS
  Participants
    Hispanic or Latino | 0 | 3 | 3 | 3 | 9
    Not Hispanic or Latino | 75 | 220 | 220 | 222 | 737
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of all patients included in the trial. Population: TS
  Participants
    American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
    Asian | 2 | 3 | 0 | 2 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 1 | 3 | 5
    White | 73 | 216 | 218 | 216 | 723
    More than one race | 0 | 2 | 4 | 3 | 9
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Pain on movement of worst procedure (POMwp) [Mean (Standard Deviation); unit: Units on scale] — Pain on movement (POM) was used to assess pain measurement for back and neck pain. The standardized movements have been established for which the measurement was taken. POMwp was the POM measure that gave the highest score at baseline; i.e. POM of worst procedure. Pain intensity was assessed at rest after standing in an upright position relatively motionless for 1 minute. The pain was evaluated by asking patient 'How would you rate your pain right now?' and by using a visual analogue scale (VAS) ranging from 0-10 cm wherein 0 cm = no pain to 10 cm = worst pain possible. Population: TS
  Units on scale | 7.20 (1.246) | 7.22 (1.157) | 7.29 (1.274) | 7.28 (1.148) | 7.26 (1.198)
Country [Number; unit: Participants] — The list of countries from which the respective number of patients had been enrolled. Population: TS
  Participants
    Germany | 69 | 205 | 205 | 205 | 684
    Russia | 6 | 18 | 18 | 20 | 62
Application site [Number; unit: Participants] — POM was assessed by patients on performance of standardized, muscle group specific movements measured using a VAS on application sites. Back and Neck were defined as application sites for this study. Acute back and neck pain was studied in this trial. Number of patients with either neck or back as an application site were presented here. Population: TS
  Participants
    Neck | 45 | 126 | 129 | 130 | 430
    Back | 30 | 97 | 94 | 95 | 316

OUTCOME MEASURES:

1. Primary Outcome: Change in POM Between Baseline and Day 2 Evening, 1 Hour After Drug Application
Description: Pain on movement (POM) was used to assess pain measurement for back and neck pain. The standardized movements have been established for which the measurement was taken. POMwp was the POM measure that gave the highest score at baseline; i.e. POM of worst procedure. Pain intensity was assessed at rest after standing in an upright position relatively motionless for 1 minute. The pain was evaluated by asking patient 'How would you rate your pain right now?' and by using a visual analogue scale (VAS) ranging from 0-10 centimeters (cm) wherein 0 cm = no pain to 10 cm = worst pain possible. The results presented here are adjusted mean change from baseline and standard error for POMwp in cm.
Time Frame: Baseline and Day 2
Population: Full analysis set (FAS): All patients in treated set with a baseline value pre application for POMwp at Visit 1 and at least 1 POMwp value during assessment times at Visit 1 (Day 1 morning 1h after application), Visit 2 (Day 2, morning 1h after application), Visit 3 (Day 2 evening before application) or Visit 3 (Day 2 evening 1h after application)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Number analyzed (Participants) | 75 | 222 | 222 | 225
Units on a scale | -2.45 (0.252) | -3.26 (0.160) | -2.33 (0.160) | -3.05 (0.159)
Statistical Analysis 1: Comparison: Placebo Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A Mixed Model Repeat Measures (MMRM) analysis was used to compare change in POMwp from baseline between placebo and combination therapy diclofenac + capsaicin. MMRM model included fixed effects of treatment, country, application site (back/neck), time and fixed covariates of baseline POMwp and baseline POMwp by time interaction; Test type: Superiority; p = 0.0303, Mixed Models Analysis; Mean Difference (Net) = -0.60, 95% CI 2-sided [-1.15 to -0.06], Standard Error of Mean 0.277 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: Capsaicin (0.075%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A Mixed Model Repeat Measures (MMRM) analysis was used to compare change in POMwp from baseline between capsaicin and combination therapy diclofenac + capsaicin. MMRM model included fixed effects of treatment, country, application site (back/neck), time and fixed covariates of baseline POMwp and baseline POMwp by time interaction; Test type: Superiority; p = 0.2886, Mixed Models Analysis; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.18 to 0.60], Standard Error of Mean 0.197 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: Diclofenac (2%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A Mixed Model Repeat Measures (MMRM) analysis was used to compare change in POMwp from baseline between diclofenac and combination therapy diclofenac + capsaicin. MMRM model included fixed effects of treatment, country, application site (back/neck), time and fixed covariates of baseline POMwp and baseline POMwp by time interaction; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = -0.72, 95% CI 2-sided [-1.10 to -0.33], Standard Error of Mean 0.197 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

2. Secondary Outcome: POMwp Area Under the Curve (AUC) Calculated From 0 to 72 Hours (h) (POMwp AUC(0-72 h))
Description: This is a key secondary endpoint. AUC for POMwp calculated from 0 to 72 h that is for first three treatment days using the trapezoidal rule divided by the observation time. The results presented here are adjusted mean and standard error for POMwp AUC (0-72 h) in centimeters (cm). The AUC represents POMwp as an average over the first 3 treatment days (Day 1 until Day 4 morning) - it is not meant here as a pharmacokinetics (PK) parameter (concentration over time).
Time Frame: 0 to 72 hours after start of treatment
Population: Treated set (TS)
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Number analyzed (Participants) | 75 | 223 | 223 | 225
cm | 4.62 (0.213) | 3.95 (0.145) | 4.81 (0.145) | 4.25 (0.143)
Statistical Analysis 1: Comparison: Placebo Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; An analysis of covariance (ANCOVA) was used to compare POMwp AUC(0-72 h) between placebo and combination therapy diclofenac + capsaicin; Test type: Superiority; p = 0.0956, ANCOVA; ANCOVA includes treatment, country, and application site (back/neck) as fixed effects, and baseline POMwp as a continuous covariate; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.80 to 0.07], Standard Error of Mean 0.221 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: Capsaicin (0.075%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; An analysis of covariance (ANCOVA) was used to compare POMwp AUC(0-72 h) between capsaicin and combination therapy diclofenac + capsaicin; Test type: Superiority; p = 0.0564, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.30, 95% CI 2-sided [-0.01 to 0.61], Standard Error of Mean 0.157 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: Diclofenac (2%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; An analysis of covariance (ANCOVA) was used to compare POMwp AUC(0-72 h) between diclofenac and combination therapy diclofenac + capsaicin; Test type: Superiority; p = 0.0004, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.56, 95% CI 2-sided [-0.87 to -0.25], Standard Error of Mean 0.157 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

3. Secondary Outcome: POMwp Area Under the Curve (AUC) Calculated From 0 to 120 Hours (h) (POMwp AUC(0-120 h))
Description: This is a key secondary endpoint. AUC for POMwp calculated from 0 to 120 h that is for first five treatment days using the trapezoidal rule divided by the observation time. The results presented here are adjusted mean and standard error for POMwp AUC (0-120 h) in centimeters (cm). The AUC represents POMwp as an average over the first 5 treatment days (Day 1 until Day 6 morning) - it is not meant here as a PK parameter (concentration over time).
Time Frame: 0 to 120 hours after start of treatment
Population: TS
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Number analyzed (Participants) | 75 | 223 | 223 | 225
cm | 3.92 (0.230) | 3.10 (0.156) | 4.10 (0.156) | 3.41 (0.154)
Statistical Analysis 1: Comparison: Placebo Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; An analysis of covariance (ANCOVA) was used to compare POMwp AUC(0-120 h) between placebo and combination therapy diclofenac + capsaicin; Test type: Superiority; p = 0.0347, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.50, 95% CI 2-sided [-0.97 to -0.04], Standard Error of Mean 0.238 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: Capsaicin (0.075%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; An analysis of covariance (ANCOVA) was used to compare POMwp AUC(0-120 h) between capsaicin and combination therapy diclofenac + capsaicin; Test type: Superiority; p = 0.0622, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.02 to 0.65], Standard Error of Mean 0.169 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: Diclofenac (2%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; An analysis of covariance (ANCOVA) was used to compare POMwp AUC(0-120 h) between diclofenac and combination therapy diclofenac + capsaicin; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.68, 95% CI 2-sided [-1.01 to -0.35], Standard Error of Mean 0.169 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

4. Secondary Outcome: Number of Patients With Decrease in POMwp of at Least 30% From Baseline
Description: This outcome measures the pattern of number of patients with a decrease in POMwp of at least 30% from baseline at 1 hour after dosing on Day 2 evening.
Time Frame: Baseline and day 2
Population: TS
Measure: Number; unit: Participants
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Number analyzed (Participants) | 75 | 223 | 223 | 225
Participants | 34 | 150 | 107 | 134
Statistical Analysis 1: Comparison: Placebo Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A logistic regression was used to compare change in number of patients with a decrease in POMwp of at least 30% from baseline between placebo and combination therapy diclofenac + capsaicin. The likelihood-ratio test was used to test for differences between treatments; Test type: Superiority; p = 0.0202, Regression, Logistic; Logistic regression model include country and application site as covariates. Odds ratio was calculated as combination treatment/individual treatment; Odds Ratio (OR) = 1.882, 95% CI 2-sided [1.10 to 3.21]
Statistical Analysis 2: Comparison: Capsaicin (0.075%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A logistic regression was used to compare change in number of patients with a decrease in POMwp of at least 30% from baseline between capsaicin and combination therapy diclofenac + capsaicin. The likelihood-ratio test was used to test for differences between treatments; Test type: Superiority; p = 0.1206, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.732, 95% CI 2-sided [0.49 to 1.09]
Statistical Analysis 3: Comparison: Diclofenac (2%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A logistic regression was used to compare change in number of patients with a decrease in POMwp of at least 30% from baseline between diclofenac and combination therapy diclofenac + capsaicin. The likelihood-ratio test was used to test for differences between treatments; Test type: Superiority; p = 0.0122, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.629, 95% CI 2-sided [1.11 to 2.39]

5. Secondary Outcome: Number of Patients With Decrease in POMwp of at Least 50% From Baseline
Description: This outcome measures the pattern of number of patients with a decrease in POMwp of at least 50% from baseline at 1 hour after dosing on Day 2 evening.
Time Frame: Baseline and day 2
Population: TS
Measure: Number; unit: Participants
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Number analyzed (Participants) | 75 | 223 | 223 | 225
Participants | 20 | 95 | 50 | 85
Statistical Analysis 1: Comparison: Placebo Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A logistic regression was used to compare change in number of patients with a decrease in POMwp of at least 50% from baseline between placebo and combination therapy diclofenac + capsaicin. The likelihood-ratio test was used to test for differences between treatments; Test type: Superiority; p = 0.0643, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.729, 95% CI 2-sided [0.97 to 3.09]
Statistical Analysis 2: Comparison: Capsaicin (0.075%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A logistic regression was used to compare change in number of patients with a decrease in POMwp of at least 50% from baseline between capsaicin and combination therapy diclofenac + capsaicin. The likelihood-ratio test was used to test for differences between treatments; Test type: Superiority; p = 0.3479, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.833, 95% CI 2-sided [0.57 to 1.22]
Statistical Analysis 3: Comparison: Diclofenac (2%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A logistic regression was used to compare change in number of patients with a decrease in POMwp of at least 50% from baseline between diclofenac and combination therapy diclofenac + capsaicin. The likelihood-ratio test was used to test for differences between treatments; Test type: Superiority; p = 0.0004, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 2.125, 95% CI 2-sided [1.40 to 3.22]

6. Secondary Outcome: Change From Baseline in POMwp (cm) at Day 6 Morning
Description: Pain on movement (POM) was used to assess pain measurement for back and neck pain. The standardized movements have been established for which the measurement was taken. POMwp was the POM measure that gave the highest score at baseline; i.e. POM of worst procedure. Pain intensity was assessed at rest after standing in an upright position relatively motionless for 1 minute. The pain was evaluated by asking patient 'How would you rate your pain right now?' and by using a visual analogue scale (VAS) ranging from 0-10 cm wherein 0 cm = no pain to 10 cm = worst pain possible. The results presented here are adjusted mean change from baseline and standard error for POMwp in centimeters (cm).
Time Frame: Baseline and Day 6
Population: TS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Number analyzed (Participants) | 75 | 223 | 223 | 225
Units on a scale | -3.83 (0.282) | -5.08 (0.175) | -3.77 (0.175) | -4.88 (0.174)
Statistical Analysis 1: Comparison: Placebo Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Mean Difference (Net) = -1.05, 95% CI 2-sided [-1.67 to -0.44], Standard Error of Mean 0.313 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: Capsaicin (0.075%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.3726, Mixed Models Analysis; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.24 to 0.64], Standard Error of Mean 0.223 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: Diclofenac (2%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -1.12, 95% CI 2-sided [-1.56 to -0.68], Standard Error of Mean 0.223 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

7. Secondary Outcome: Change From Baseline in Pressure Algometry (PA) at Day 2 Evening, Before Drug Application
Description: PA is a method described to determine pressure pain threshold (PPT) by applying controlled pressure to a given body point. The results presented here are adjusted mean change from baseline and standard error for PA.
Time Frame: Baseline and Day 2
Population: TS
Measure: Least Squares Mean (Standard Error); unit: Newton/centimeter square (N/cm^2)
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Number analyzed (Participants) | 75 | 223 | 223 | 225
Newton/centimeter square (N/cm^2) | 3.89 (0.795) | 3.46 (0.526) | 3.00 (0.530) | 3.77 (0.526)
Statistical Analysis 1: Comparison: Placebo Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A Mixed Model Repeat Measures (MMRM) analysis was used to compare change in PA from baseline between placebo and combination therapy diclofenac + capsaicin. MMRM model included fixed effects of treatment, country, application site (back/neck), time and fixed covariates of baseline PA and baseline PA by time interaction; Test type: Superiority; p = 0.8810, Mixed Models Analysis; Mean Difference (Net) = -0.13, 95% CI 2-sided [-1.78 to 1.53], Standard Error of Mean 0.844 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: Capsaicin (0.075%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A Mixed Model Repeat Measures (MMRM) analysis was used to compare change in PA from baseline between capsaicin and combination therapy diclofenac + capsaicin. MMRM model included fixed effects of treatment, country, application site (back/neck), time and fixed covariates of baseline PA and baseline PA by time interaction; Test type: Superiority; p = 0.6094, Mixed Models Analysis; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.87 to 1.49], Standard Error of Mean 0.601 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: Diclofenac (2%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; A Mixed Model Repeat Measures (MMRM) analysis was used to compare change in PA from baseline between diclofenac and combination therapy diclofenac + capsaicin. MMRM model included fixed effects of treatment, country, application site (back/neck), time and fixed covariates of baseline PA and baseline PA by time interaction; Test type: Superiority; p = 0.2047, Mixed Models Analysis; Mean Difference (Net) = 0.76, 95% CI 2-sided [-0.42 to 1.95], Standard Error of Mean 0.602 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

8. Secondary Outcome: Change From Baseline in Pressure Algometry (PA) at Day 6 Morning
Description: as for outcome 7
Time Frame: Baseline and Day 6
Population: TS
Measure: Least Squares Mean (Standard Error); unit: Newton/centimeter square (N/cm^2)
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
Number analyzed (Participants) | 75 | 223 | 223 | 225
Newton/centimeter square (N/cm^2) | 8.01 (1.199) | 9.38 (0.737) | 7.64 (0.740) | 9.66 (0.737)
Statistical Analysis 1: Comparison: Placebo Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.2193, Mixed Models Analysis; Mean Difference (Net) = 1.65, 95% CI 2-sided [-0.98 to 4.27], Standard Error of Mean 1.339 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: Capsaicin (0.075%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.7672, Mixed Models Analysis; Mean Difference (Net) = 0.28, 95% CI 2-sided [-1.58 to 2.15], Standard Error of Mean 0.949 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: Diclofenac (2%) Gel vs Diclofenac (2%) +Capsaicin (0.075%) Gel; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.0339, Mixed Models Analysis; Mean Difference (Net) = 2.02, 95% CI 2-sided [0.15 to 3.88], Standard Error of Mean 0.950 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

ADVERSE EVENTS:
Time Frame: From first drug administration until 2 days after the last drug administration, i.e. up to 8 days.
Description: An adverse event (AE) was defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product. The event did not necessarily have to have a causal relationship with this treatment. TS (as treated) has been used for assessment of AEs.
Arm/Group | Placebo Gel | Capsaicin (0.075%) Gel | Diclofenac (2%) Gel | Diclofenac (2%) +Capsaicin (0.075%) Gel
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/223 | 0/223 | 0/225
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/223 | 0/223 | 0/225
Other Adverse Events (participants affected / at risk) | 4/75 | 29/223 | 7/223 | 26/225
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Gel (N=75) | Capsaicin (0.075%) Gel (N=223) | Diclofenac (2%) Gel (N=223) | Diclofenac (2%) +Capsaicin (0.075%) Gel (N=225)
Burning sensation (General disorders) | 0 | 16 | 1 | 12
Nasopharyngitis (Infections and infestations) | 4 | 9 | 4 | 3
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 7 | 2 | 12

LIMITATIONS AND CAVEATS:
A possible limitation of this study design related to the warming effect that is attributable to the topical application of capsaicin, which could potentially have led to inadvertent unblinding of treatment assignments in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT02700815/SAP_000.pdf
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT02700815/Prot_001.pdf